CLINICAL TRIAL: NCT07155603
Title: Visual Aids for Colonoscopy Preparation: A Prospective Study on Patient Understanding and Bowel Cleanliness in Colonoscopy Patients
Acronym: VACP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Prof. Dr. med. Jörg Daniel Leuppi, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-01572
Record Dates: First submitted 2025-03-10; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: The Effect of Audio-visual Aids on Bowel Cleanliness; Audiovisual Aids

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Consent (Control Group) (Active Comparator): The traditional informed consent process involves the provision of written documents and verbal explanation to the patient regarding the colonoscopy procedure, risks, and preparation requirements
  Interventions: Behavioral: Animated Video Group 1
- Animated Video 1 (Experimental): Patients of this group will be asked to watch the Visikon animated videos, in addition to receiving standard informed consent
  Interventions: Behavioral: Animated Video Group 1

INTERVENTIONS:
Behavioral: Animated Video Group 1 — The animated video intervention provides a clear and engaging multimedia explanation of the colonoscopy procedure in multiple languages. It includes visual aids to help explain the process, preparation instructions, risks, and expected outcomes, aiming to improve patient comprehension and adherence.

SUMMARY:
Effective communication in healthcare is critical for improving patient outcomes, particularly in enhancing health literacy and enabling informed decision-making. Traditional informed consent for colonoscopy often fails to clearly explain the procedure, risks, and preparation requirements, leading to inadequate bowel preparation, longer procedures, and missed lesions. Standard educational materials like videos and written instructions are often impersonal, lack cultural inclusivity, and fail to engage patients effectively. Emerging tools, such as the multilingual, visually enhanced Meine Behandlung video series from Visikon®, aim to improve patient comprehension and adherence. This study seeks to compare the effectiveness of these animated videos against traditional consent methods in enhancing patient understanding and adherence, particularly for complex procedures like colonoscopy, which is crucial for diagnosing and preventing colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scheduled for a routine outpatient colonoscopy procedure
* Capable of understanding communication in German and willing to participate in the study

Exclusion Criteria:

* Patients with cognitive impairments
* Those unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Bowel Preperation | 24 months
  The objective of assessing the primary endpoint the patient's bowel cleanliness, will be measured during the routine colonoscopy, using the Boston Bowel Preperation Scale.
  The Boston Bowel Preparation Scale (BBPS) is a validated tool used to assess the cleanliness of the colon during a colonoscopy,
  Each of the three segments of the colon (right, transverse, and left) is assigned a score ranging from 0 to 3, with the following criteria:
  Total Score 0: The entire colon is unprepared, and no mucosa is visible. Total Score 1-3: Poor preparation, significant portions of the mucosa are not visible.
  Total Score 4-6: Fair preparation, with some portions of the mucosa visible but others obscured.
  Total Score 7-9: Good to excellent preparation, with most or all mucosa well visualized.
  Interpretation Scores of 0-3: Generally considered inadequate for proper assessment and diagnosis, likely requiring repeat preparation and examination.
  Scores of 4-6: Indicative of suboptimal preparation

SECONDARY OUTCOMES:
Patient Health Literacy & Communication Satisfaction | 24 months
  The secondary outcome seeks to assess the patient's health literacy and general communication satisfaction. This will be done by assessing their answers to the Health Literacy Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital of Baselland, Liestal, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided